CLINICAL TRIAL: NCT06902922
Title: Impact of Severe Tricuspid Regurgitation Correction on Gut Microbiota and Gastrointestinal Function
Acronym: Tri-GuM
Status: Not yet recruiting | Type: Observational
Sponsor: Francesco Maisano (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Francesco Maisano, Head of Cardiac Surgery Department; Director of the Heart Valve Center, IRCCS Ospedale San Raffaele
Organization: IRCCS Ospedale San Raffaele (Other)
Other Study IDs: Tri-GuM
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Tricuspid Regurgitation (TR)
Keywords: tricuspid regurgitation; gut microbiota; gastrointestinal; heart; heart valve disease; tricuspid valve disease; transcatheter; T-TEER
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- T-TEER: Adult patients, able to sign the Informed Consent Form, with TR ≥ severe who will be treated with T-TEER

SUMMARY:
Tricuspid regurgitation (TR) is gaining increasing attention within the cardiological community due to its poor prognosis, challenging clinical presentation and difficult treatment.

TR causes decreased forward cardiac output and increased intravascular pressure upstream, which lead to peripheral oedema, ascites, hepatic congestion and kidney failure.

The microbiota is also getting increasing attention and changes in microbiota have been already associated with cardiovascular disease.

The impact of hemodynamic effects of TR on the gut microbiota however is still unknown.

Patients affected by TR frequently complain abdominal distension and anorexia. We hypothesize that, due to increased venous congestion, TR may induce impaired gut function with modification in the microbiota and that TR correction may induce reverse changes.

This study will enroll patients treated with Transcatheter Tricuspid Edge-to-Edge Repair (T-TEER) at the Valve Center of San Raffaele Hospital due to severe TR.

In addition to the standard of care, before T-TEER, for all patients 2 additional blood samples, 1 urine and 1 fecal sample will be collected.

3 months after the procedure, all patients will be re-assessed at the Valve Center outpatient clinic as standard of care. At this stage for all patients 2 blood samples, 1 urine and 1 fecal sample will be collected again for the purpose of the study. The microbiota metabolites of patients after 3 months from the procedure will be compared to those at baseline according to the degrees of residual TR.

To assess the reproducibility of the microbiota results and to explore an intrinsic short-term variation in microbiome composition within single patients, a subgroup of 30 patients will undergo a low intervention substudy repeating the measurements (2 blood, 1 urine and 1 fecal) within 10 days, both at baseline and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, able to sign the Informed Consent Form, admitted to OSR Heart Valve Center with TR ≥ severe treated with T-TEER.

Exclusion Criteria:

* Concomitant ≥ severe MR. Such patients may be treated with M-TEER and be re-evaluated after 3 months: if TR is ≥ severe and MR is ≤ moderate the patient may then be enrolled.
* Surgical candidates
* Recent < 6 months cardiac coronary or structural procedure
* CAD requiring intervention
* other valvular disease > moderate
* Treatment with transcatheter tricuspid replacement
* Age <18 years
* Inability or unwillingness to sign informed consent
* Kidney dialysis
* Acute infection
* Inflammatory bowel diseases
* Gastrointestinal diseases
* Previous gastrointestinal surgery
* Active cancer
* Active autoimmune or inflammatory diseases
* Treatments with antibiotics or probiotics within one month
* Emergency procedures
* Patients enrolled in interventional studies that may confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with TR ≥ severe who will undergo T-TEER
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiota Changes | 3 months
  The microbiota metabolites production in patients affected by severe TR and their changes after transcatheter TR correction will be measured at 3-months, compared to baseline, in terms of c differential abundance in microbiota metabolites, according to residual TR groups

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No